CLINICAL TRIAL: NCT04359992
Title: Study of Hemostasis in Case of Severe COVID-19
Acronym: THROMBOVID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7774
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Extra blood sample — 3 extra blood samples at day 0, 2 and 7

SUMMARY:
The COVID-19 outbreak has led to a significant increase in the number of patients admitted to intensive care for respiratory distress. Early data indicate a particularly high risk of thrombotic risk to viral lung disease, particularly in the most severe patients, with a particularly high incidence of pulmonary embolism. Catheter thrombosis and extra-renal purification filters are also abnormally common. These thrombotic complications could contribute to the mortality observed in this pathology. The introduction of early curative anticoagulation in the most severe patients has just been proposed by the perioperative hemostasis interest group

Biologically, a significant proportion of patients hospitalized in intensive care have a marked biological inflammatory syndrome, associated with signs of activation of clotting (a frank increase in D-dimers). The presence of circulating anticoagulants is common. Interestingly, thrombocytosis, normally observed in such inflammatory syndromes, is absent.

In this context, it seems legitimate to explore these patients from a hemostasis perspective to identify the factors that cause this thrombotic over-risk, in order to minimize the occurrence of these complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (<18y)
* With a SARS-CoV-2 infection confirmed by RT-PCR
* Hospitalized in intensive care

Exclusion Criteria:

* Patients under guardianship/curator
* Anemia at 7 g/dL at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in intensive care for severe COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-17 (Estimated); Primary Completion 2021-04-17 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Platelet activation intensity with the occurrence of clinical thrombotic complications | Change of platelet activity from admission's day in intensive care unit to 2 days and 7 days

REFERENCES:
- [Derived] Tacquard C, Mouriaux C, Delabranche X, Bourdon C, Eckly A, Magnenat S, Sattler L, Gachet C, Mertes PM, Hechler B, Mangin PH. Platelet dysfunction and thrombus instability in flow conditions in patients with severe COVID-19. Thromb Res. 2023 Jan;221:137-148. doi: 10.1016/j.thromres.2022.11.004. Epub 2022 Nov 8. PMID 36376109